CLINICAL TRIAL: NCT06851884
Title: Efficacité d'Interventions Pour améliorer le vécu Des Proches de Patients hospitalisés en réanimation. RELIEF, un Essai Plateforme
Brief Title: Effectiveness of Informational and Educational Tools to Improve the Experience of Relatives of ICU Patients. RELIEF, a Platform Trial
Acronym: RELIEF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP240666
Record Dates: First submitted 2025-02-10; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-01

CONDITIONS: Post Traumatic Stress Disorder PTSD
MeSH Terms: conditions — Combat Disorders | interventions — Standard of Care; Videotape Recording

STUDY DESIGN:
Intervention Model Description: Randomized platform trial designed to investigate a clinical question across multiple subpopulations and involving multiple interventions.
  The trials integrated into the platform trial are randomized and may be either conventional trials or adaptive MAMS (Multi-Arms Multi-Stage) trials. These involve multiple arms and phases, allowing for the adaptive evaluation of several interventions, with the possibility of adding or removing interventions during the trial.
  Additionally, the trials include a hybrid control arm that combines randomized concurrent controls and historical external controls from an observational cohort.
  Trial 1 : randomization according to a 1:2:2:2 ratio into one of the 4 arms:
  * Control
  * Video capsules
  * Comic strips
  * Virtual reality
  Trial 2 : randomization according to a 1:2 ratio into the control or intervention arm (set of "end-of-life and grief" informational and educational tools, including a video capsule, a cartoon, and a kit of 2 leaflets).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Trial 1 : Control (Active Comparator): Standard care with universal welcome leaflet. The control group is a hybrid, also including historical external controls from the cohort "Syndrome de Stress Post-traumatique chez les Proches de Patients Admitted to the Intensive Care Unit: A Multicentric, Observational, Prospective Study" according to the center's usual practice
  Interventions: Other: Standard of Care (SOC)
- Trial 1 : Video Capsule arm (Experimental)
  Interventions: Other: Video capsules
- Trial 1 : Cartoon arm (Experimental)
  Interventions: Other: Cartoon
- Trial 1 : Virtual reality arm (Experimental)
  Interventions: Other: Virtual reality
- Trial 2 : Control (Active Comparator): Standard care with universal welcome leaflet. The control group is a hybrid, also including historical external controls from the cohort "Syndrome de Stress Post-traumatique chez les Proches de Patients Admitted to the Intensive Care Unit: A Multicentric, Observational, Prospective Study" according to the center's usual practice
  Interventions: Other: Standard of Care (SOC)
- Trial 2 : set of "end-of-life and grief" informational and educational tools (Experimental)
  Interventions: Other: Set of "end-of-life and grief" informational and educational tools

INTERVENTIONS:
Other: Standard of Care (SOC) — Universal welcome leaflet on patient admission
  Arms: Trial 1 : Control
Other: Video capsules — 3 video capsules of 3 minutes each
  Arms: Trial 1 : Video Capsule arm
Other: Cartoon — 3 cartoons
  Arms: Trial 1 : Cartoon arm
Other: Virtual reality — 3 virtual reality programs
  Arms: Trial 1 : Virtual reality arm
Other: Set of "end-of-life and grief" informational and educational tools — Including a video capsule, a cartoon, and a kit of two leaflets
  Arms: Trial 2 : set of "end-of-life and grief" informational and educational tools
Other: Standard of Care (SOC) — Universal welcome leaflet on patient admission
  Arms: Trial 2 : Control

SUMMARY:
The admission of a patient to an intensive care unit (ICU) is associated with high levels of acute stress, anxiety, and depression among relatives, as well as extreme emotions such as fear, guilt, distress, and helplessness. In addition to these emotions, relatives also struggle to understand the information provided by the medical team-only half of the information is fully understood. These emotional and cognitive difficulties can become obstacles in decision-making processes and may have medium- and long-term consequences on their psychological well-being, particularly in terms of post-traumatic stress disorder (PTSD), anxiety, and depression. Three months after the patient is discharged from the ICU, one-third of relatives exhibit symptoms of PTSD.

The aim of this research is to propose a variety of informational and educational tools to improve relatives' understanding of both the ICU context and the information provided, with the goal of reducing the risk of developing PTSD in the months following the patient's discharge or death.

ELIGIBILITY:
Inclusion Criteria:

Trial 1 :

Relatives of patients with the following characteristics: ≥18 years old, treated in intensive care with invasive mechanical ventilation for at least 48 hours having received a visit from at least one relative within the first 72 hours.

* ≥18 years old
* Identified, if possible, by the patient as the reference person or person to be informed, or, if the patient is unable to communicate, identified by the healthcare providers as the "patient's reference relative."
* Understanding and speaking French • Having provided their phone contact information Only one relative of the patient is included in the study.

Trial 2 :

Relatives of patients with the following characteristics: ≥18 years old, having been treated in intensive care with invasive mechanical ventilation for at least 48 hours, for whom a decision of withhold or withdraw treatment has been made with expected death in intensive care.

* ≥18 years old
* Identified, if possible, by the patient as the reference person or person to be informed, or, if the patient is unable to communicate, identified by healthcare providers as the "patient's reference relative."
* Present at the end-of-life conference (announcement of the EOL decision)
* Understanding and speaking French
* Having provided their phone contact information

Only one relative of the patient is included in the study. They are included just before or just after the end-of-life conference.

Exclusion Criteria:

Patients :

* Planned or considered organ donation
* Detained or deprived of liberty
* Under guardianship or curatorship
* No social security

Relatives :

* Social context making follow-up and telephone interviews difficult (homeless individuals, not residing in Europe or the overseas territories)
* Inability to provide a "stable" personal mobile number (temporary phone number or not in their own name or the name of their spouse/partner)
* Under guardianship or curatorship
* Inability to communicate by phone (hearing impairments, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 562 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Post-Traumatic Stress Disorder (PTSD) | At 3 months
  Assessed with PCL-5 scale three months after the patient's discharge or death. The PCL-5 scale, Post-traumatic stress disorder CheckList version DSM-5 (PCL-5) [PCL-5, 8/14/2013, Weathers, Litz, Keane, Palmieri, Marx, & Schnurr - National Center for PTSD] includes 20 items addressing PTSD symptoms according to DSM-5 criteria. Each item is rated from 0 ("not at all") to 4 ("extremely") for a total score between 0 and 80).

SECONDARY OUTCOMES:
Trial 1 : Measure the impact of each of the 3 sets of tools on the overall understanding of relatives in intensive care | Up to 6 months
  Measure the impact of each of the 3 sets of informational and educational tools on the overall understanding of relatives in intensive care (diagnosis, prognosis, treatment) at the time of discharge from intensive care (questionnaire)
Trial 1 : Measure the impact of each of the 3 sets of tools on the anxiety and depression symptoms of relatives | Up to 6 months
  Measure the impact of each of the 3 sets of informational and educational tools on the anxiety and depression symptoms of relatives at the time of discharge from intensive care (HADS scale).
  HADS is a self-administered scale of 14 items which assessed levels of depression and anxiety, divided into 2 subscales of 7 items (Anxiety or HADS-A, Depression or HADS-D). Each item is scored on a scale of 0 to 3. A score is generated for each of the two sub-scales (sum of the 7 items, ranging from 0 to 21). Limit scores, for each of the scores, distinguish: non-cases or asymptomatic ones (score ≤ 7); probable or borderline cases (score 8-10); clearly or clinically symptomatic cases (score ≥ 11).
Trial 1 & 2 : Sleep quality of relatives | At inclusion
  Evaluated by ISI : Insomnia Severity Index It is a 7 questions scale. Each question is rated on a scale from 0 to 4, with 0 indicating no problems and 4 indicating very severe problems. The total score can range from 0 to 28, with higher scores indicating more severe insomnia.
Trial 1 & 2 : Sleep quality of relatives | At 3 months
  Evaluated by ISI : Insomnia Severity Index It is a 7 questions scale. Each question is rated on a scale from 0 to 4, with 0 indicating no problems and 4 indicating very severe problems. The total score can range from 0 to 28, with higher scores indicating more severe insomnia.
Trial 1 & 2 : Sleep quality of relatives | At 6 months
  Evaluated by ISI : Insomnia Severity Index It is a 7 questions scale. Each question is rated on a scale from 0 to 4, with 0 indicating no problems and 4 indicating very severe problems. The total score can range from 0 to 28, with higher scores indicating more severe insomnia.
Trial 1 & 2 : Symptoms of post-traumatic dissociation | At inclusion
  Evaluated by PDEQ : Post-traumatic Dissociation Questionnaire. Total score ranges from 0 to 48. The higher the score the more severe the dissociation symptoms are.
Trial 1 & 2 : satisfaction of relatives regarding communication with the intensive care teams | At 3 months
  Satisfaction assessed on a 8-step scale regarding communication with intensive care team
Trial 1 & 2 Post-traumatic stress disorder | At 6 months
  Trial 1 : Measure the impact of each of the 3 sets of informational and educational tools on the risk of developing post-traumatic stress disorder Trial 2 : Measure the impact of EOL of informational and educational tools on the risk of developing post-traumatic stress disorder
  Assessed with PCL-5 scale six months after the patient's discharge or death. The PCL-5 scale, Post-traumatic stress disorder CheckList version DSM-5 (PCL-5) [PCL-5, 8/14/2013, Weathers, Litz, Keane, Palmieri, Marx, & Schnurr - National Center for PTSD] includes 20 items addressing PTSD symptoms according to DSM-5 criteria. Each item is rated from 0 ("not at all") to 4 ("extremely") for a total score between 0 and 80).
  6 months after the patient's discharge or death
Trial 1 & 2 : anxiety and depression symptoms of relatives | At 3 months
  Trial 1 : Measure the impact of each of the 3 sets of informational and educational tools on the risk of developing anxiety and depression symptoms in relatives
  Trial 2 : Measure the impact of EOL informational and educational tools on the risk of developing anxiety and depression symptoms in relatives
  HADS is a self-administered scale of 14 items which assessed levels of depression and anxiety, divided into 2 subscales of 7 items (Anxiety or HADS-A, Depression or HADS-D). Each item is scored on a scale of 0 to 3. A score is generated for each of the two sub-scales (sum of the 7 items, ranging from 0 to 21). Limit scores, for each of the scores, distinguish: non-cases or asymptomatic ones (score ≤ 7); probable or borderline cases (score 8-10); clearly or clinically symptomatic cases (score ≥ 11).
  3 months after the patient's discharge or death
Trial 1 & 2 : anxiety and depression symptoms of relatives | At 6 months
  Trial 1 : Measure the impact of each of the 3 sets of informational and educational tools on the risk of developing anxiety and depression symptoms in relatives
  Trial 2 : Measure the impact of EOL informational and educational tools on the risk of developing anxiety and depression symptoms in relatives
  HADS is a self-administered scale of 14 items which assessed levels of depression and anxiety, divided into 2 subscales of 7 items (Anxiety or HADS-A, Depression or HADS-D). Each item is scored on a scale of 0 to 3. A score is generated for each of the two sub-scales (sum of the 7 items, ranging from 0 to 21). Limit scores, for each of the scores, distinguish: non-cases or asymptomatic ones (score ≤ 7); probable or borderline cases (score 8-10); clearly or clinically symptomatic cases (score ≥ 11).
  6 months after the patient's discharge or death
Trial 1 & 2 : Past traumatic experiences | At 3 months
  Trauma History Screen (THS) The THS typically asks individuals to respond to a series of yes/no questions about whether they've experienced specific types of trauma. They include : Physical abuse, Sexual abuse, Witnessing violence, Accidents or natural disasters, Military combat, Emotional abuse, Neglect.
  The score is the number of traumatic events.
Trial 1 & 2 : Risk of developing prolonged grief 6 months after the patient's death | At 6 months
  Trial 1 : Measure, in bereaved relatives, the impact of informational and educational tools on the risk of developing prolonged grief
  Trial 2 : Measure the impact of EOL informational and educational tools on the risk of developing prolonged grief
  Prolonged Grief Disorder Scale PG-13 The score ranges from 0 to 52. Total scores of 30 or above generally indicate that the individual may be experiencing Prolonged Grief Disorder (PGD) and should be considered for further evaluation.
  Lower scores suggest that the individual is not experiencing clinically significant prolonged grief symptom
Trial 1 & 2 : Consumption of medical care and acts by relatives | At inclusion
  Using MEDEC tool (medical care consumption and acts) It summarizes frequency and type of care
Trial 1 & 2 : Consumption of medical care and acts by relatives | Up to 6 months
  Using MEDEC tool (medical care consumption and acts) It summarizes frequency and type of care
  During the 6 months following the patient's discharge or death
Trial 1&2 : Feasability of use of the tool | Up to 6 months
  Trial 1 : Percentage of care provider who were able to hand over the 3 sets of informational and educational tools to the patient's relatives, as well as their satisfaction
  Trial 2 : Percentage of care provider who wereable to hand over the EOL informational and educational tools to the patient's relatives, as well as their satisfaction
Trial 1 & 2 : Quality of tools assessed by families by a self-assessment questionnaire | At 3 months
  self-assessment questionnaire with 14 items

IPD SHARING:
Plan to Share IPD: Undecided